CLINICAL TRIAL: NCT01813500
Title: Host Immune Response to Clostridium Difficile Infection in Inflammatory Bowel Disease Patients
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Collaborators: Cepheid (Industry); Optimer Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Principal Investigator, Francis Farraye, MD, Principal Investigator, Boston Medical Center
Other Study IDs: H-31226
Record Dates: First submitted 2013-03-15; First posted 2013-03-19 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Crohn's Disease; Ulcerative Colitis; Clostridium Difficile; Inflammatory Bowel Disease
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, stool
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IBD Patients: Subjects with Crohn's Disease or Ulcerative colitis. IBD patients will be asked to provide a blood and stool sample.
  Interventions: Other: Blood and stool sample
- Control Subjects: Subjects without Crohn's Disease or Ulcerative Colitis. Controls will also be asked to provide a blood and stool sample.
  Interventions: Other: Blood and stool sample

INTERVENTIONS:
Other: Blood and stool sample — Subjects are asked to provide a blood sample (6 to 10cc) and a stool sample. An additional blood sample will be requested if the subject has a flare.

SUMMARY:
The inflammatory bowel diseases (IBD), ulcerative colitis (UC) and Crohn's disease (CD) are chronic conditions affecting approximately 1.4 million Americans. The burden of Clostridium difficile infection (CDI), a frequent cause of infectious diarrhea is mediated by toxins A and B and is increasing faster in IBD patients, than the general population. Clinically, CDI in patients with IBD leads to a range of clinical syndromes from symptomless carriage, to severe life threatening colitis, colectomy and death.

This pilot study will look at the relationship between IBD and this variable host immune response. Clostridium difficile colonization (asymptomatic carrier state) is lower in the IBD population than in the general population. In the general population, high antitoxin titers have been linked with colonization and low antitoxin titers with recurrent disease. The investigators hypothesize that patients with IBD will have a lower Clostridium difficile colonization and will have lower antibody titers than the control group. Additionally those with lower titers will have an increased risk of developing CDI.

In Aim 1 the investigators will determine Clostridium colonization in IBD subjects by stool study (including CD, UC and UC patients after IPAA) compared to non-IBD subjects (controls). In Aim 2 the investigators will compare antitoxin titers in these IBD subjects compared to controls. In Aim 3 the investigators will follow these subjects for 12 months and calculate the incidence of CDI in patients with IBD compared to controls and associations with anti-toxin titers.

DETAILED DESCRIPTION:
This is a two part pilot study, with the initial phase (Aim 1 and Aim 2) being a cross-sectional epidemiological analysis of Clostridium difficile colonization and anti-toxin antibodies in the IBD population compared to non-IBD patients.

The second phase (Aim 3) is a pilot nested case-control study that will follow both groups of patients prospectively for 12 months to see who develops either colonization or active CDI and correlate these to clinical demographics and serum Clostridium difficile anti-toxin antibodies.

All subjects age eighteen and older who are able to give consent, have a diagnosis of inflammatory bowel disease (see clinical definition of IBD below) and are followed in the Center for Digestive Disease (CDD) are eligible for this study. Control subjects will also be followed in the CDD without a diagnosis of IBD. All subjects will be recruited from routine scheduled visits when seen as outpatients at the CDD or will be identified from the inpatient Gastroenterology consult service or at the Internal Medicine Department at Shapiro as part of Dr. Qazi's rotation(see recruitment section).

Subjects will be recruited in a block fashion to minimize confounding variables and ensure groups with equal amount of diarrhea and to keep a 3:1 ratio of IBD to controls. Subject will be recruited on a consecutive basis in a block of 32 slots. Within that block, 8 slots will be for the control group (4 with diarrhea, 4 without) and 24 IBD patients (12 with diarrhea, 12 without). Once all slots are filled then the next block will begin.

For Aim 1 and Aim 2: Upon enrollment subjects from both groups will provide blood and stool samples (details of amount and timing discussed below) and a retrospective chart review will document pre-determined data (as listed below). Total time requirement upon enrollment would be about 10-15 minutes.

For Aim 3: This is an intention-to-treat analysis; control subjects who become diagnosed with IBD during the study period will be kept in the control group. Patients will be followed for a 12 month period:

If during that time there is no CDI then there will be no further study visits, only data review at the end of the study period.

If a subject develops diarrhea in either group, treatment will be per standard of care (detailed below) and research team will be alerted by primary Gastroenterologist or GI consult team. If deemed appropriate by clinical team stool will be sent for C diff (per SOC) and if positive, then repeat blood samples for anti-toxin titers may be collected (for research purposes). At the end of the 12 month study period data will be reviewed.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects must be 18 years of age or older, able to provide written informed consent, and able to comply with the requirements of the study.
2. All subjects must speak English. Non-English subjects are not included because of lack of funding for interpreter services and clinical resources could not be used for research purposes.
3. For Control Group only: Non-IBD subject seen in CDD during routine visit or on inpatient consult service
4. For IBD Group Only: Chart history of IBD (either UC or CD) confirmed by colonoscopy, pathology or gastroenterology clinical judgment

Exclusion Criteria:

1. Any subject planning on moving out of the area in the next year
2. Any patient not able to give informed consent
3. Any subject unwilling or not able to give stool sample upon enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with Crohn's Disease and Ulcerative Colitis or healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Colonization | 12 Months
  Determine Clostridium colonization in IBD patients during clinical remission and during flares (including CD, UC and UC patients after IPAA) compared to controls

SECONDARY OUTCOMES:
Incidence | 12 months
  Determine the incidence of CDI in patients with IBD (including CD, UC and UC patients after IPAA) compared to controls and correlate to anti-toxin titer levels using the methods as outlined above

CONTACTS AND LOCATIONS:
Overall Officials: Francis A Farraye, MD, Principal Investigator — Boston Medical Center Department of Gastroenterology
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Berg AM, Kelly CP, Farraye FA. Clostridium difficile infection in the inflammatory bowel disease patient. Inflamm Bowel Dis. 2013 Jan;19(1):194-204. doi: 10.1002/ibd.22964. PMID 22508484